CLINICAL TRIAL: NCT01641822
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study of Aztreonam for Inhalation Solution (AZLI) in a Continuous Alternating Therapy (CAT) Regimen of Inhaled Antibiotics for the Treatment of Chronic Pulmonary Pseudomonas Aeruginosa Infection in Subjects With Cystic Fibrosis
Brief Title: Phase 3 Study of Aztreonam for Inhalation Solution (AZLI) in a Continuous Alternating Therapy Regimen for the Treatment of Chronic Pseudomonas Aeruginosa Infection in Patients With CF
Acronym: AZLI CAT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-205-0170; 2015-000398-11 (EudraCT Number)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Results first posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Aztreonam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AZLI (Active Comparator): Participants will be randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens: AZLI for 28 days followed by TIS for 28 days.
  Interventions: Drug: AZLI; Drug: Tobramycin inhalation solution
- Placebo (Placebo Comparator): Participants will be randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens: placebo to match AZLI for 28 days followed by TIS for 28 days.
  Interventions: Drug: Placebo to match AZLI; Drug: Tobramycin inhalation solution

INTERVENTIONS:
Drug: AZLI — Aztreonam for Inhalation Solution (AZLI) 75 mg 3 times daily combined with diluent administered using an eFlow nebulizer
  Other Names: Cayston®
  Arms: AZLI
Drug: Placebo to match AZLI — Placebo to match AZLI 3 times daily combined with diluent administered using an eFlow nebulizer
  Arms: Placebo
Drug: Tobramycin inhalation solution — Tobramycin inhalation solution (TIS) 300 mg 2 times daily using a PARI® LC Plus nebulizer and DeVilbiss Pulmo-Aide® air compressor
  Other Names: TOBI®

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of a CAT regimen with aztreonam for inhalation solution (AZLI) and tobramycin inhalation solution (TIS) in adult and pediatric subjects with cystic fibrosis (CF) and pulmonary Pseudomonas aeruginosa (PA) infection. Participants will be enrolled in a 28 day TIS run-in phase, and will be eligible for randomization in the comparative phase if they have not received non-study oral antibiotics for a respiratory event, or IV or inhaled antibiotics for any indication between Visits 2 and 3, have not developed a condition requiring hospitalization or other change in clinical status which, in the opinion of the investigator would preclude their ability to continue in the study, and have demonstrated at least 50% TIS compliance. Participants enrolled in the comparative phase will be randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens: AZLI or placebo for 28 days followed by TIS for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of CF
* Presence of PA in 2 lower respiratory tract cultures in the 12 months prior to screening
* Forced expiratory volume (FEV)1 ≥ 25 and ≤ 75% predicted
* History of 1 hospitalization or 1 course of IV antibiotics for an acute respiratory exacerbation in the 12 months prior to screening

Exclusion Criteria:

* Concurrent use of oral, IV or inhaled antibiotics at enrollment
* Concurrent hospitalization at enrollment
* History of local or systemic hypersensitivity to monobactams or aminoglycoside antibiotics or history of aminoglycoside antibiotic associated toxicity

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-12; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bresnik, MD, Study Director — Gilead Sciences
Locations (71):
- United States (71):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - University of California - San Diego, La Jolla, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Kaiser Permanente Medical Center, Oakland, California
  - National Jewish Health, Denver, Colorado
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Central Florida Pulmonary Group, Altamonte Springs, Florida
  - University of Florida, Gainesville, Florida
  - South Broward Hospital dba Memorial Healthcare System, Hollywood, Florida
  - Nemours Children's Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami, Miami, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Nemour's Children's Clinic, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - Tampa General Hospital, Tampa, Florida
  - Emory Cystic Fibrosis Center, Atlanta, Georgia
  - Georgia Health, Augusta, Georgia
  - St. Lukes Medical Center, Boise, Idaho
  - University of Chicago, Chicago, Illinois
  - Chicago CF Care Specialists NFP dba Cystic Fibrosis Institure, Glenview, Illinois
  - Indiana University, Indianapolis, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Maine Medical Center, Portland, Maine
  - Boston Children's Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Spectrum Health - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St. Louis University - Cardinal Glennon Children's Hospital, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Children's Lung Specialists, Las Vegas, Nevada
  - Dartmouth Hitchcock Specialty Care Clinic, Bedford, New Hampshire
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Morristown Medical Center, Morristown, New Jersey
  - UNM Clinical and Translational Center, Albuquerque, New Mexico
  - Albany Medical College, Albany, New York
  - Long Island Jewish Medical Center - Adult CF & Bronchiectasis Center, New Hyde Park, New York
  - Gunnar Esiason Adult CF and Lung Program, New York, New York
  - SUNY Upstate University, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Akron Children's Hospital, Akron, Ohio
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - UC Health - University of Cincinnati, Cincinnati, Ohio
  - The Toledo Hospital/Toledo Children's Hospital CF Center, Toledo, Ohio
  - OU Health Sciences Center, Oklahoma City, Oklahoma
  - Santiago Reyes, MD, Oklahoma City, Oklahoma
  - Geisinger Clinic, Danville, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Children's Foundation Research Institute/UTHSC, Memphis, Tennessee
  - Vanderbilt Children's Hospital, Nashville, Tennessee
  - Austin Children's Chest Associates, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Alamo Clinical Research Associates, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - Vermont Lung Center at the University of Vermont, Colchester, Vermont
  - University of Virginia, Charlottesville, Virginia
  - Children's Hospital of the King's Daughters, Norfolk, Virginia
  - VCU Children's Hospital, Richmond, Virginia
  - West Virginia University, Morgantown, West Virginia
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Flume PA, Clancy JP, Retsch-Bogart GZ, Tullis DE, Bresnik M, Derchak PA, Lewis SA, Ramsey BW. Continuous alternating inhaled antibiotics for chronic pseudomonal infection in cystic fibrosis. J Cyst Fibros. 2016 Nov;15(6):809-815. doi: 10.1016/j.jcf.2016.05.001. Epub 2016 May 24. PMID 27233377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in the United States. The first participant was screened on 13 December 2012. The last study visit occurred on 15 January 2015.
Pre-assignment Details: Following enrollment, participants received tobramycin inhalation solution (TIS) in the TIS Run-In Phase, and if still eligible were randomized 1 to 1 to receive aztreonam for inhalation solution (AZLI) or placebo to match AZLI alternating with TIS in the Comparative Phase.
Groups:
- TIS Run-In Treatment Group: Enrolled participants received 28 days of TIS (300 mg 2 times daily) during the run-in phase.
- AZLI: Participants were randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens AZLI (75 mg 3 times daily) for 28 days followed by TIS (300 mg 2 times daily) for 28 days.
- Placebo: Participants were randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens: placebo to match AZLI for 28 days followed by TIS (300 mg 2 times daily) for 28 days.
Period: Run-in Phase
Arm/Group | TIS Run-In Treatment Group | AZLI | Placebo
Started | 107 | 0 | 0
Completed | 93 (3 participants who completed the TIS Run-In Phase did not continue to the Comparative Phase.) | 0 | 0
Not Completed | 14 | 0 | 0
Not completed — Noncompliance with study drug | 1 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0
Not completed — Withdrew consent | 1 | 0 | 0
Not completed — Protocol-specified criteria for withdraw | 9 | 0 | 0
Period: Comparative Phase
Arm/Group | TIS Run-In Treatment Group | AZLI | Placebo
Started | 0 (Participants continuing into the Comparative Phase were randomized to the AZLI or Placebo group.) | 43 | 47
Received Randomized Study Drug Treatment | 0 | 42 | 46
Completed | 0 | 37 | 37
Not Completed | 0 | 6 | 10
Not completed — Noncompliance with study drug | 0 | 1 | 0
Not completed — Investigator's discretion | 0 | 0 | 1
Not completed — Pregnancy | 0 | 0 | 1
Not completed — Adverse event, serious fatal | 0 | 1 | 0
Not completed — Withdrew consent | 0 | 3 | 7
Not completed — Protocol-specified criteria for withdraw | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Analysis Set: all randomized participants
Groups:
- AZLI: Participants were randomized to receive 3 cycles of treatment, each cycle consisting alternating regimens: AZLI (75 mg 3 times daily) for 28 days followed by TIS (300 mg 2 times daily) for 28 days.
- Total: Total of all reporting groups
Arm/Group | AZLI | Placebo | Total
Number analyzed (Participants) | 43 | 47 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (12.10) | 28.0 (10.88) | 28.4 (11.42)
Age, Customized [Number; unit: participants]
  6 - 12 years | 3 | 1 | 4
  13 - 17 years | 5 | 6 | 11
  ≥ 18 years | 35 | 40 | 75
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 28 | 52
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 4 | 9
  Not Hispanic or Latino | 38 | 43 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 | 1
  White | 41 | 45 | 86
  Other | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 43 | 47 | 90
FEV1 % predicted at Day 1 [Mean (Standard Deviation); unit: percentage of FEV1 % predicted] — Forced expiratory volume (FEV)1 is defined as the maximal volume of air that can be exhaled in 1 second. FEV1 % predicted is defined as FEV1 of the participant divided by the average FEV1 in the population for any person of similar age, sex, race, and body composition.
  percentage of FEV1 % predicted | 49.95 (17.500) | 50.25 (15.131) | 50.11 (16.213)
CFQ-R Respiratory Score at Day 1 [Mean (Standard Deviation); unit: units on a scale] — Respiratory symptoms (eg, coughing, congestion, wheezing) were assessed with the Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS). The range of scores (units) was 0 to 100 with higher scores indicating fewer symptoms.
  units on a scale | 59.72 (18.408) | 64.24 (15.044) | 62.11 (16.773)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Protocol-defined Exacerbations (PDE) From Baseline Through Week 24
Description: PDEs were characterized by a change or worsening from baseline of 1 or more documented signs or symptoms (decreased exercise tolerance, increased cough, increased sputum or chest congestion, decreased appetite, or other signs or symptoms) associated with the use of non-study IV or inhaled antibiotics and be verified by a blinded independent adjudication committee.
Time Frame: Baseline in the comparative phase to the end of study (average time on study during the Comparative Phase: 155.4 days)
Population: Intent-to-Treat (ITT) Analysis Set: all randomized participants
Measure: Number; unit: PDEs per participant year
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 43 | 47
PDEs per participant year | 1.309 | 1.762
Statistical Analysis 1: Comparison: AZLI vs Placebo; Ratio between rates; Test type: Superiority or Other; p = 0.25, Negative binomial regression; Risk Ratio (RR) = 0.743, 95% CI 2-sided [0.446 to 1.238]

2. Secondary Outcome: Average Actual Change From Baseline in FEV1 % Predicted Across All Courses of AZLI/Placebo Treatment (Weeks 4, 12 and 20)
Description: FEV1 % predicted is defined as FEV1 of the patient divided by the average FEV1 in the population for any person of similar age, sex and body composition. The adjusted mean is from a mixed-effect model repeated measures (MMRM) analysis. The model includes terms for baseline value, previous exacerbations (1, 2, ≥ 3), treatment, visit (categorical), and treatment by visit interaction.
Time Frame: Comparative Phase: Baseline and Weeks 4, 12 and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Error); unit: percentage of FEV1 % predicted
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 42 | 45
percentage of FEV1 % predicted | 1.37 (0.674) | 0.04 (0.658)
Statistical Analysis 1: Comparison: AZLI vs Placebo; Difference in change in FEV1 % predicted; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis — The p-value is from an MMRM analysis. The model includes terms for baseline value, previous exacerbations (1, 2, ≥ 3), treatment, visit (categorical), and treatment by visit interaction; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-0.55 to 3.2]

3. Secondary Outcome: Percentage of Participants Who Used Non-study IV or Inhaled Antibiotics for PDEs
Time Frame: Baseline in the comparative phase to the end of study (average time on study during the Comparative Phase: 155.4 days)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 43 | 47
percentage of participants | 48.8 | 55.3
Statistical Analysis 1: Comparison: AZLI vs Placebo; Comparison of percentages; Test type: Superiority or Other; p = 0.67, Fisher Exact

4. Secondary Outcome: Time to First Protocol-defined Pulmonary Exacerbation
Description: The time to first protocol-defined pulmonary exacerbation was calculated using the Kaplan-Meier method.
Time Frame: Baseline in the comparative phase to the end of study (average time on study during the Comparative Phase: 155.4 days)
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 43 | 47
days | 175 [76.0 to NA] — Not reached due to an insufficient number of events | 140.0 [90.0 to NA] — Not reached due to an insufficient number of events
Statistical Analysis 1: Comparison: AZLI vs Placebo; Comparison of time to exacerbation; Test type: Superiority or Other; p = 0.71, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.50 to 1.59]

5. Secondary Outcome: Rate of Hospitalizations for a Respiratory Event
Description: The rate of hospitalizations for a respiratory event per participant year was calculated using negative binomial regression analysis.
Time Frame: Baseline in the comparative phase to the end of study (average time on study during the Comparative Phase: 155.4 days)
Population: ITT Analysis Set
Measure: Number; unit: hospitalizations per participant year
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 43 | 47
hospitalizations per participant year | 1.043 | 1.624
Statistical Analysis 1: Comparison: AZLI vs Placebo; Comparison of hospitalization rate; Test type: Superiority or Other; p = 0.14, Negative binomial regression; Risk Ratio (RR) = 0.642, 95% CI 2-sided [0.355 to 1.164]

6. Secondary Outcome: Average Change From Baseline in the CFQ-R Respiratory Symptom Scale (RSS) Score Across All Courses of AZLI/Placebo Treatment (Weeks 4, 12 and 20)
Description: Respiratory symptoms (eg, coughing, congestion, wheezing) were assessed with the Cystic Fibrosis Questionnaire - Revised (CFQ-R) Respiratory Symptoms Scale (RSS). The range of scores (units) was 0 to 100 with higher scores indicating fewer symptoms. The adjusted mean is from a mixed-effect model repeated measures (MMRM) analysis. The model includes terms for baseline value, previous exacerbations (1, 2, ≥ 3), treatment, visit (categorical), and treatment by visit interaction.
Time Frame: Comparative Phase: Baseline and Weeks 4, 12 and 20
Population: Participants in the ITT Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AZLI | Placebo
Number analyzed (Participants) | 39 | 45
units on a scale | 1.00 (1.736) | -2.06 (1.629)
Statistical Analysis 1: Comparison: AZLI vs Placebo; Difference in change in CFQ-R RSS; Test type: Superiority or Other; p = 0.21, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]; Mean Difference (Final Values) = 3.06, 95% CI 2-sided [-1.71 to 7.82]

ADVERSE EVENTS:
Time Frame: TIS Run-In Treatment Group: up to 28 days (plus 30 days if not continuing to the comparative phase). Comparative phase: from first dose of AZLI or Placebo through 30 days after last dose (average 155.4 days).
Description: Safety analysis set: participants who were enrolled and received at least 1 dose of study drug
Arm/Group | TIS Run-In Treatment Group | AZLI | Placebo
Serious Adverse Events (participants affected / at risk) | 4/107 | 21/42 | 24/46
Other Adverse Events (participants affected / at risk) | 27/107 | 38/42 | 44/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TIS Run-In Treatment Group (N=107) | AZLI (N=42) | Placebo (N=46)
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 | 0
Blindness unilateral (Eye disorders) | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 3
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 0 | 1
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 2 | 9 | 5
Pneumonia (Infections and infestations) | 1 | 1 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 | 1 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 9 | 13
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TIS Run-In Treatment Group (N=107) | AZLI (N=42) | Placebo (N=46)
Abdominal pain (Gastrointestinal disorders) | 0 | 4 | 1
Constipation (Gastrointestinal disorders) | 0 | 4 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 5
Nausea (Gastrointestinal disorders) | 0 | 6 | 10
Vomiting (Gastrointestinal disorders) | 0 | 5 | 9
Chest discomfort (General disorders) | 7 | 8 | 13
Chest pain (General disorders) | 0 | 4 | 7
Chills (General disorders) | 0 | 3 | 5
Exercise tolerance decreased (General disorders) | 0 | 3 | 12
Fatigue (General disorders) | 6 | 11 | 17
Pyrexia (General disorders) | 0 | 8 | 13
Forced expiratory volume decreased (Investigations) | 0 | 4 | 2
Pulmonary function test decreased (Investigations) | 0 | 11 | 10
Weight decreased (Investigations) | 0 | 4 | 5
Decreased appetite (Metabolism and nutrition disorders) | 0 | 5 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 3 | 4
Headache (Nervous system disorders) | 0 | 7 | 8
Sinus headache (Nervous system disorders) | 0 | 3 | 2
Anxiety (Psychiatric disorders) | 0 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 21 | 32 | 33
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 13 | 24
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 11
Increased viscosity of bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 5
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 11 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 8
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 7
Sputum discoloured (Respiratory, thoracic and mediastinal disorders) | 0 | 5 | 3
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 12 | 20 | 31
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 6 | 9 | 9
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 4 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years